CLINICAL TRIAL: NCT00332072
Title: Safety and Efficacy Study of Bimatoprost/Timolol Fixed Combination in Patients Wtih Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-021T
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension | interventions — Bimatoprost

INTERVENTIONS:
Drug: bimatoprost/timolol fixed combination

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Bimatoprost/Timolol Fixed Combination in the treatment of glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension or chronic glaucoma in both eyes
* Patient needs IOP-lowering drug in both eyes

Exclusion Criteria:

* Uncontrolled medical condition
* Contraindication to beta-adrenoceptor antagonist therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2001-08; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
IOP

CONTACTS AND LOCATIONS:
Locations (1):
- Ogden, Utah, United States

REFERENCES:
- [Derived] Lewis RA, Gross RL, Sall KN, Schiffman RM, Liu CC, Batoosingh AL; Ganfort Investigators Group II. The safety and efficacy of bimatoprost/timolol fixed combination: a 1-year double-masked, randomized parallel comparison to its individual components in patients with glaucoma or ocular hypertension. J Glaucoma. 2010 Aug;19(6):424-6. doi: 10.1097/IJG.0b013e3181bdb586. No abstract available. PMID 19855289